CLINICAL TRIAL: NCT02746653
Title: Effectiveness and Safety of Gordian Surgical's TroClose1200™, a Trocar With built-in Closure Device Capability, in Subjects Undergoing Laparoscopic Surgery
Brief Title: Effectiveness and Safety of Gordian Surgical's TroClose1200™
Acronym: GOR-CLN-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gordian Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOR-CLN-01
Record Dates: First submitted 2016-04-12; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Hernia
Keywords: Fascia Closure Device, hernia,
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of TroClose1200(TM) for access port and closure device (Experimental): TroClose in 1 port
  Interventions: Device: TroClose1200(TM)

INTERVENTIONS:
Device: TroClose1200(TM) — Creation of access port and closure it by the same device, TroClose1200(TM)

SUMMARY:
The use of the TroClose1200™ will be done in at least one 12mm planned access port per the TroClose1200™ Instruction for Use. The procedure will be performed routinely. Adverse Events and device malfunctions, if any, will be recorded. Subjects will be hospitalized in accordance with the hospital guidance. All subjects will be followed at 2 weeks (+/- 4 days), at 6 weeks (+/- 1 week), at 12 months (+/- 1 month) and at 24 months (+/- 2 months) in which healing, signs of hernia and adverse events will be recorded. In the 12 and 24 months visit, the hernia signs will be evaluated by ultrasound.

DETAILED DESCRIPTION:
Subjects that sign the Informed Consent Form will be evaluated for eligible for the study per eligibility criteria. Subject medical background and underlying disease requiring intervention will be taken at screening. Procedure will be scheduled. Subjects that will eventually, for any reason, will not be operated with the TroClose1200™, will be considered as "screen failures". The use of the TroClose1200™ will be done in at least one 12mm planned access port per the TroClose1200™ Instruction for Use. The procedure will be performed routinely. Duration of use of the TroClose1200™ each time it is used will be measured, as well as the entire procedure duration, and the type of procedure. Adverse Events and device malfunctions, if any, will be recorded. The video seen in the monitors during the procedure will be kept as source data for any further analysis. The location of the TroClose1200™ used, as well as the other trocars used location, will be drawn on a special chart. Subjects will be hospitalized in accordance with the hospital guidance. All subjects will be followed at 2 weeks (+/- 4 days), at 6 weeks (+/- 1 week), at 12 months (+/- 1 month) and at 24 months (+/- 2 months) in which healing, signs of hernia and adverse events will be recorded. In the 12 and 24 months visit, the hernia signs will be evaluated by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old and less than 65 years.
2. Subject is a candidate for laparoscopic surgery with at least one 12 mm trocar is to be used apart from the endoscopic access port.
3. Subject is capable and willing to comply with, and be present at, the follow-up clinic visits of the 6 weeks visit.
4. Subject is able and willing to sign a written informed consent form.

Exclusion Criteria:

1. Patients presenting factors that affect the scarring process, such as malnutrition (serum proteins <5 g/dl or Albumin below 3 g/dl).
2. Advanced cancer.
3. Perioperative hemodynamic instability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome is the proportion of successfully created ports and their closure by the TRoClosed | Perioperative
  Operator will record trocar insertion, anchor deployment, ability to accommodate laparoscopic surgical tools within the cannula and closure ability of the port for each of the ports created by the TroClose

SECONDARY OUTCOMES:
Secondary efficacy outcome assessed by hernia signs at 6,12,and 24 months | Up to 2 years
  Hernia signs assessment by palpation by the surgeon at 6 weeks. Hernia signs assessment by palpation by the surgeon and by US at 12 months. Hernia signs assessment by palpation by the surgeon and by US at 24 months.
Secondary Safety Outcome assessed by surgical complications | up to 6 weeks
  Surgical complication by Clavien Dindo classification perioperatively and at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hagar Mizrahi, Dr., Principal Investigator — Poryia Medical Center, Israel
Locations (1):
- Poryia Medical Center, Teberias, Israel